CLINICAL TRIAL: NCT00377858
Title: Comparison of Two Approaches to Basal-Bolus Insulin Therapy in Patients With Type 2 Diabetes and Inadequate Glycemic Control on Oral Therapy: Comparison of Premixed Insulin Lispro Mid Mixture With Separate Basal and Bolus Insulin Injections
Brief Title: Comparison of Two Approaches to Insulin Therapy in Patients With Type 2 Diabetes (IOOX)
Acronym: IOOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10936; F3Z-MC-IOOX
Record Dates: First submitted 2006-09-11; First posted 2006-09-19 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro Mid Mixture (Experimental): Insulin lispro mid mixture (MM) up to three times a day (TID)
  Interventions: Drug: Insulin lispro mid mixture (MM)
- Insulin Glargine (Active Comparator): Insulin glargine daily with insulin lispro at mealtime (up to 3 injections) as needed.
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin lispro mid mixture (MM) — Patient specific adjusted dose, three times a day (TID), subcutaneous (SC) injection x 36 weeks
  Other Names: Humalog; Mid Mix
  Arms: Insulin Lispro Mid Mixture
Drug: Insulin glargine — Patient specific adjusted dose, every day (QD), subcutaneous (SC) injection x 36 weeks
  Arms: Insulin Glargine

SUMMARY:
A study of patients with type 2 diabetes and inadequate glycemic control on two or more oral antihyperglycemic agents comparing adding insulin lispro mid mixture to the oral antihyperglycemic agents to adding insulin glargine to the oral antihyperglycemic agents.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Have been receiving oral antihyperglycemic medications (OAM) without insulin including at least two of the following at maximally tolerated doses, AND meet the minimum dosing criteria shown: Metformin 1500 mg/day, Sulfonylurea 1/2 the maximum daily dose, according to package insert, Thiazolidinedione (TZD) 30 mg/day pioglitazone or 4 mg/day rosiglitazone. The OAMs also must be used in accordance with the product label
* Have a hemoglobin A1c greater than or equal to 7.5% and less than or equal to 12.0%.

Exclusion Criteria:

* Are taking a TZD dose greater than what is indicated in combination with insulin according to the TZD label.
* Are taking any other glucose-lowering agents not mentioned in Inclusion Criterion.
* Have taken acarbose, miglitol, pramlintide, exenatide, repaglinide, or nateglinide in the past 6 weeks or for a total of 30 days or more in the last 24 weeks.
* Have a body mass index greater than 40 kg/m2.
* Have had more than one episode of severe hypoglycemia in the last24 weeks
* Are pregnant, intend to be pregnant during the course of the study or are breastfeeding
* Have clinically significant cardiac, renal, hematologic, oncologic, or hepatic disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fitzroy, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremantle, Western Australia
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granby, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regina, Saskatchewan
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mantes-la-Jolie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Menton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-Si/Kyunggi-Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Almería
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilbao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga

REFERENCES:
- [Derived] Hayes RP, Curtis B, Ilag L, Nelson DR, Wong M, Funnell M. Expectations about insulin therapy, perceived insulin-delivery system social acceptability, and insulin treatment satisfaction contribute to decreases in insulin therapy self-efficacy in patients with type 2 diabetes after 36 weeks insulin therapy. J Diabetes. 2013 Sep;5(3):358-67. doi: 10.1111/1753-0407.12037. Epub 2013 May 28. PMID 23489710
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 636 patients were screened; 128 were screen failures; 24 discontinued prior to randomization; 484 patients were randomized. Baseline Characteristics are provided for the Intent to Treat Population, which was defined as patients with baseline and at least one post-baseline value.
Period: Overall Study
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Started | 242 | 242
Had at Least One Post-Baseline Value | 239 | 240
Completed | 211 | 215
Not Completed | 31 | 27
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Lost to Follow-up | 6 | 1
Not completed — Physician Decision | 5 | 5
Not completed — Protocol Violation | 3 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Entry Criteria Not Met | 2 | 0
Not completed — Sponsor Decision | 1 | 2
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine | Total
Number analyzed (Participants) | 239 | 240 | 479
Age Continuous [Mean (Standard Deviation); unit: years] | 58.40 (9.21) | 59.45 (9.87) | 58.92 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 120 | 251
  Male | 108 | 120 | 228
Region of Enrollment [Number; unit: participants]
  Australia | 18 | 19 | 37
  Canada | 27 | 24 | 51
  France | 21 | 19 | 40
  Greece | 19 | 20 | 39
  India | 26 | 29 | 55
  Korea, Republic of | 24 | 25 | 49
  Mexico | 51 | 47 | 98
  Russian Federation | 24 | 26 | 50
  Spain | 29 | 31 | 60
Body Mass Index (BMI) Group [Number; unit: participants] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  participants
    BMI <25 kg/m^2 | 34 | 48 | 82
    BMI ≥25 kg/m^2 and <30 kg/m^2 | 106 | 103 | 209
    BMI ≥30 kg/m^2 | 99 | 89 | 188
Duration of Diabetes Group [Number; unit: participants]
  <5 years | 28 | 27 | 55
  ≥5 years and ≤10 years | 95 | 100 | 195
  >10 years | 116 | 113 | 229
Hemoglobin A1c (HbA1c) Group [Number; unit: participants]
  ≤8.5% HbA1c | 60 | 67 | 127
  >8.5% HbA1c | 179 | 173 | 352
Race/Ethnicity [Number; unit: participants]
  African | 2 | 1 | 3
  Caucasian | 134 | 136 | 270
  East Asian | 25 | 27 | 52
  Hispanic | 51 | 46 | 97
  West Asian (Indian sub-continent) | 27 | 30 | 57
Body Height [Mean (Standard Deviation); unit: centimeters (cm)] | 163.27 (9.27) | 164.68 (9.48) | 163.98 (9.39)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 29.51 (4.76) | 29.00 (4.55) | 29.25 (4.66)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 78.85 (15.50) | 78.87 (15.10) | 78.86 (15.28)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 10.86 (5.54) | 11.79 (7.29) | 11.33 (6.48)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent HbA1c] | 9.55 (1.18) | 9.39 (1.17) | 9.47 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) at 36 Week Endpoint
Description: Level of hemoglobin A1c at endpoint.
Time Frame: 36 weeks
Population: Number of participants in the per-protocol population. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percent HbA1c
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 188 | 195
percent HbA1c | 7.66 (0.37) | 7.49 (0.36)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Assuming 15% drop-out rate after randomization, remaining 213 patients in each treatment group would allow confirmation of noninferiority with no treatment difference and a noninferiority limit of 0.3% using upper limit of 2-sided confidence interval at significance level of 0.05 with 80% power; Test type: Non-Inferiority or Equivalence — Noninferiority margin of 0.3% based on prior studies indicating an HbA1c difference of 0.6% in patients treated with lispro and sulfonylurea compared with those treated with sulfonylurea and metformin; p = 0.097, ANCOVA; ANCOVA Model: Variable=Treatment + Baseline HbA1c Stratum + Sulfonylurea stratum + Country + Baseline HbA1c Stratum; Mean Difference (Net) = 0.17, 95% CI [-0.03 to 0.37] — The two-sided 95% confidence interval of the Least Squares Mean difference between the two treatments is for (Insulin Lispro Mid Mixture minus Insulin Glargine)

2. Secondary Outcome: Hemoglobin A1c (HbA1c) at Interval Visits
Description: Levels of HbA1c at 12 weeks and 24 weeks and 36 weeks.
Time Frame: 12, 24, and 36 weeks
Population: Number of randomized patients with baseline and at least one post-baseline value. Intent to treat population.
Measure: Least Squares Mean (Standard Error); unit: percent HbA1c
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 222 | 222
percent HbA1c
  12 Week Interval (n=222, n=222) | 8.02 (0.32) | 7.85 (0.31)
  24 Week Interval (n=206, n=217) | 7.53 (0.33) | 7.36 (0.32)
  36 Week Interval (n=202, n=208) | 7.53 (0.37) | 7.44 (0.37)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.047, ANCOVA — P-value for 12 Week Interval; ANCOVA Model: Variable=Treatment + Baseline HbA1c + Baseline HbA1c stratum + Sulfonylurea stratum + Country; Mean Difference (Net) = 0.16, 95% CI [0.00 to 0.33] — The two-sided 95% confidence interval of the Least Squares Mean difference between the two treatments is for Insulin Lispro Mid Mix minus Insulin Glargine
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.043, ANCOVA — P-value for 24 Week Interval; ANCOVA Model: Variable=Treatment + Baseline HbA1c + Baseline HbA1c stratum + Sulfonylurea stratum + Country; Mean Difference (Net) = 0.18, 95% CI [0.01 to 0.35] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.343, ANCOVA — P-value for 36 Week Interval; ANCOVA Model: Variable=Treatment + Baseline HbA1c + Baseline HbA1c stratum + Sulfonylurea stratum + Country; Mean Difference (Net) = 0.10, 95% CI [-0.10 to 0.29] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Patients Who Achieved Hemoglobin A1c Less Than or Equal to 6.5%, Greater Than 6.5%, Less Than 7%, Greater Than or Equal to 7%, Less Than or Equal to 7%, and Greater Than 7% at Interval Visits and Endpoint
Time Frame: 12-24-36 weeks
Population: Number of randomized patients with baseline and at least one post-baseline value. Intent to treat population. If the patient completed the trial, the endpoint was 36 weeks (Week 36), but if the patient dropped out of the study early, the last observation carried forward (LOCF) was considered as the endpoint (Endpoint).
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 234 | 235
percentage of participants
  Week 12: HbA1c ≤7.0% (n=222, n=222) | 21.2 | 25.2
  Week 12: HbA1c >7.0% (n=222, n=222) | 78.8 | 74.8
  Week 12: HbA1c <7.0% (n=222, n=222) | 18.9 | 21.6
  Week 12: HbA1c ≥7.0% (n=222, n=222) | 81.1 | 78.4
  Week 12: HbA1c ≤6.5% (n=222, n=222) | 8.1 | 10.8
  Week 12: HbA1c >6.5% (n=222, n=222) | 91.9 | 89.2
  Week 24: HbA1c ≤7.0% (n=206, n=217) | 39.8 | 47.0
  Week 24: HbA1c >7.0% (n=206, n=217) | 60.2 | 53.0
  Week 24: HbA1c <7.0% (n=206, n=217) | 35.4 | 38.7
  Week 24: HbA1c ≥7.0% (n=206, n=217) | 64.6 | 61.3
  Week 24: HbA1c ≤6.5% (n=206, n=217) | 16.0 | 21.7
  Week 24: HbA1c >6.5% (n=206, n=217) | 84.0 | 78.3
  Week 36: HbA1c ≤7.0% (n=202, n=208) | 39.6 | 44.7
  Week 36: HbA1c >7.0% (n=202, n=208) | 60.4 | 55.3
  Week 36: HbA1c <7.0% (n=202, n=208) | 37.6 | 40.4
  Week 36: HbA1c ≥7.0% (n=202, n=208) | 62.4 | 59.6
  Week 36: HbA1c ≤6.5% (n=202, n=208) | 15.3 | 19.2
  Week 36: HbA1c >6.5% (n=202, n=208) | 84.7 | 80.8
  Endpoint (LOCF): HbA1c ≤7.0% (n=234, n=235) | 36.8 | 43.0
  Endpoint (LOCF): HbA1c >7.0% (n=234, n=235) | 63.2 | 57.0
  Endpoint (LOCF): HbA1c <7.0% (n=234, n=235) | 35.0 | 39.1
  Endpoint (LOCF): HbA1c ≥7.0% (n=234, n=235) | 65.0 | 60.9
  Endpoint (LOCF): HbA1c ≤6.5% (n=234, n=235) | 13.2 | 19.1
  Endpoint (LOCF): HbA1c >6.5% (n=234, n=235) | 86.8 | 80.9
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.432, Regression, Logistic — P-value for Week 12: HbA1c ≤7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.602, Regression, Logistic — P-value for 12 Week: HbA1c <7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.370, Regression, Logistic — P-value for 12 Week: HbA1c ≤6.5%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 4: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.198, Regression, Logistic — P-value for 24 Week: HbA1c ≤7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 5: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.636, Regression, Logistic — P-value for 24 Week: HbA1c <7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 6: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.185, Regression, Logistic — P-value for 24 Week: HbA1c ≤6.5%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 7: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.393, Regression, Logistic — P-value for 36 Week: HbA1c ≤7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 8: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.739, Regression, Logistic — P-value for 36 Week: HbA1c <7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 9: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.396, Regression, Logistic — P-value for 36 Week: HbA1c ≤6.5%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 10: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.227, Regression, Logistic — P-value for Endpoint (LOCF): HbA1c ≤7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 11: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.482, Regression, Logistic — P-value for Endpoint (LOCF): HbA1c <7.0%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum
Statistical Analysis 12: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.108, Regression, Logistic — P-value for Endpoint (LOCF): HbA1c ≤6.5%; Logistic Regression Model: Variable=Treatment + Baseline HbA1c + Country + Sulfonylurea Stratum

4. Secondary Outcome: 7-point Self-monitored Blood Glucose Profiles
Description: Actual daily mean blood glucose levels at specified time points.
Time Frame: Baseline, 12-24-36 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimoles per Liter (mmol/L)
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
millimoles per Liter (mmol/L)
  Baseline: Morning Pre-Meal (n=228, n=231) | 10.22 (0.91) | 9.64 (0.90)
  Baseline: Morning Postprandial Meal (n=213, n=222) | 12.49 (1.18) | 12.39 (1.16)
  Baseline: Midday Pre-Meal (n=227, n=230) | 10.15 (1.07) | 9.62 (1.05)
  Baseline: Midday Postprandial Meal (n=215, n=223) | 11.40 (1.12) | 11.22 (1.10)
  Baseline: Evening Pre-Meal (n=227, n=229) | 10.38 (1.09) | 10.31 (1.07)
  Baseline: Evening Postprandial Meal (n=226,n= 229) | 11.87 (1.05) | 11.76 (1.03)
  Baseline: 0300 Hours (n=205, n=202) | 9.37 (1.08) | 9.17 (1.06)
  12 Week: Morning Pre-Meal (n=218, n=226) | 7.26 (0.64) | 6.68 (0.63)
  12 Week: Morning Postprandial Meal (n=192, n=206) | 11.56 (0.94) | 11.28 (0.92)
  12 Week: Midday Pre-Meal (n=215, n=220) | 8.63 (0.76) | 8.10 (0.75)
  12 Week: Midday Postprandial Meal (n=196, n=209) | 9.92 (0.91) | 9.43 (0.89)
  12 Week: Evening Pre-Meal (n=216, n=221) | 8.75 (0.80) | 7.98 (0.79)
  12 Week: Evening Postprandial Meal (n=213, n= 223) | 8.23 (0.90) | 9.40 (0.89)
  12 Week: 0300 Hours (n=185, n=187) | 6.97 (0.79) | 7.12 (0.78)
  24 Week: Morning Pre-Meal (n=210, n=213) | 6.72 (0.64) | 6.07 (0.63)
  24 Week: Morning Postprandial Meal (n=193, n=201) | 9.87 (0.91) | 9.45 (0.89)
  24 Week: Midday Pre-Meal (n=209, n=213) | 7.99 (0.79) | 7.82 (0.77)
  24 Week: Midday Postprandial Meal (n=196, n=203) | 9.38 (0.90) | 9.15 (0.88)
  24 Week: Evening Pre-Meal (n=209, n=211) | 7.50 (0.81) | 6.94 (0.79)
  24 Week: Evening Postprandial Meal (n=207, n= 207) | 8.21 (0.82) | 8.69 (0.81)
  24 Week: 0300 Hours (n=181, n=184) | 7.14 (0.71) | 7.18 (0.70)
  36 Week: Morning Pre-Meal (n=200, n=210) | 6.96 (0.67) | 6.48 (0.65)
  36 Week: Morning Postprandial Meal (n=179, n=194) | 10.09 (0.92) | 10.29 (0.90)
  36 Week: Midday Pre-Meal (n=199, n=210) | 7.33 (0.77) | 7.46 (0.76)
  36 Week: Midday Postprandial Meal (n=182, n=195) | 10.31 (0.92) | 10.30 (0.91)
  36 Week: Evening Pre-Meal (n=199, n=207) | 8.13 (0.81) | 7.97 (0.79)
  36 Week: Evening Postprandial Meal (n=195, n= 225) | 9.46 (0.85) | 9.85 (0.83)
  36 Week: 0300 Hours (n=167, n=177) | 8.18 (1.06) | 8.25 (1.05)
  Endpoint: Morning Pre-Meal (n=228, n=231) | 6.98 (0.68) | 6.53 (0.67)
  Endpoint: Morning Postprandial Meal (n=213, n=222) | 9.98 (0.94) | 10.29 (0.92)
  Endpoint: Midday Pre-Meal (n=227, n=230) | 7.36 (0.80) | 7.52 (0.79)
  Endpoint: Midday Postprandial Meal (n=215, n=223) | 10.28 (0.91) | 10.34 (0.90)
  Endpoint: Evening Pre-Meal (n=227, n=229) | 8.15 (0.81) | 7.98 (0.80)
  Endpoint: Evening Postprandial Meal (n=226,n= 229) | 9.27 (0.85) | 9.84 (0.83)
  Endpoint: 0300 Hours (n=205, n=202) | 7.78 (0.75) | 7.89 (0.74)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.014, ANOVA — P-value for Baseline: Morning Pre-Meal; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.58, 95% CI [0.12 to 1.04] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.735, ANOVA — P-value for Baseline: Morning Postprandial Meal; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.11, 95% CI [-0.51 to 0.72] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.051, ANOVA — P-value for Baseline: Midday Pre-Meal; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.54, 95% CI [-0.00 to 1.08] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.536, ANOVA — P-value for Baseline: Midday Postprandial Meal; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.18, 95% CI [-0.39 to 0.75] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.793, ANOVA — P-value for Baseline: Evening Pre-Meal; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.07, 95% CI [-0.48 to 0.62] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.693, ANOVA — P-value for Baseline: Evening Postprandial Meal; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.11, 95% CI [-0.43 to 0.64] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.499, ANOVA — P-value for Baseline: 0300 Hours; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.20, 95% CI [-0.38 to 0.77] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for 12 Week: Morning Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.59, 95% CI [0.26 to 0.92] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.278, ANCOVA — P-value for 12 Week: Morning Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.28, 95% CI [-0.22 to 0.78] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value for 12 Week: Midday Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.53, 95% CI [0.14 to 0.93] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.049, ANCOVA — P-value for 12 Week: Midday Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.49, 95% CI [0.00 to 0.97] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for 12 Week: Evening Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.77, 95% CI [0.35 to 1.18] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for 12 Week: Evening Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -1.17, 95% CI [-1.63 to -0.70] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.506, ANCOVA — P-value for 12 Week: 0300 Hours; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.15, 95% CI [-0.59 to 0.29] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for 24 Week: Morning Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.65, 95% CI [0.31 to 0.99] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.094, ANCOVA — P-value for 24 Week: Morning Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.42, 95% CI [-0.07 to 0.91] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.408, ANCOVA — P-value for 24 Week: Midday Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.17, 95% CI [-0.24 to 0.59] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.351, ANCOVA — P-value for 24 Week: Midday Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.23, 95% CI [-0.25 to 0.71] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value for 24 Week: Evening Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.56, 95% CI [0.13 to 0.98] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value for 24 Week: Evening Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.48, 95% CI [-0.92 to -0.05] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.816, ANCOVA — P-value for 24 Week: 0300 Hours; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.05, 95% CI [-0.45 to 0.35] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value for 36 Week: Morning Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.49, 95% CI [0.13 to 0.85] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.438, ANCOVA — P-value for 36 Week: Morning Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.20, 95% CI [-0.71 to 0.31] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.548, ANCOVA — P-value for 36 Week: Midday Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.13, 95% CI [-0.54 to 0.29] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.964, ANCOVA — P-value for 36 Week: Midday Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.01, 95% CI [-0.50 to 0.52] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 26: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.453, ANCOVA — P-value for 36 Week: Evening Pre-Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.16, 95% CI [-0.27 to 0.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 27: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.096, ANCOVA — P-value for 36 Week: Evening Postprandial Meal; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.39, 95% CI [-0.84 to 0.07] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 28: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.770, ANCOVA — P-value for 36 Week: 0300 Hours; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.07, 95% CI [-0.51 to 0.37] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 29: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value for Endpoint: Morning Pre-Meal. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.45, 95% CI [0.11 to 0.80] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 30: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.201, ANCOVA — P-value for Endpoint: Morning Postprandial Meal. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.31, 95% CI [-0.80 to 0.17] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 31: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.430, ANCOVA — P-value for Endpoint: Midday Pre-Meal. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.16, 95% CI [-0.57 to 0.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 32: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.814, ANCOVA — P-value for Endpoint: Midday Postprandial Meal. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.06, 95% CI [-0.52 to 0.41] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 33: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.427, ANCOVA — P-value for Endpoint: Evening Pre-Meal. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.17, 95% CI [-0.24 to 0.57] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 34: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value for Endpoint: Evening Postprandial Meal. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.57, 95% CI [-1.00 to -0.14] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 35: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.569, ANCOVA — P-value for Endpoint: 0300 Hours. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.12, 95% CI [-0.51 to 0.28] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Glycemic Variability
Description: Glycemic variability was measured by mean blood glucose value (M-value), which was the mean of the intra-days self-monitoring blood glucose values, and by the mean of daily difference (MODD), which was the mean of the between-days self-monitored blood glucose values.
Time Frame: Baseline, 12-24-36 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
millimoles per liter (mmol/L)
  Baseline MODD (n=226, n=229) | 2.09 (0.33) | 2.07 (0.32)
  Baseline M-Value (n=228, n=231) | 48.02 (14.73) | 46.75 (14.47)
  12 Week MODD (n=214, n=221) | 1.51 (0.31) | 1.54 (0.31)
  12 Week M-Value (n=218, n=226) | 30.07 (7.24) | 28.49 (7.12)
  24 Week MODD (n=208, n=211) | 1.57 (0.33) | 1.66 (0.32)
  24 Week M-Value (n=210, n=213) | 22.67 (7.05) | 20.14 (6.93)
  36 Week MODD (n=198, n=206) | 1.55 (0.32) | 1.60 (0.32)
  36 Week M-Value (n=200, n=210) | 26.46 (7.26) | 27.41 (7.12)
  Endpoint MODD (n=226, n=229) | 1.51 (0.32) | 1.61 (0.31)
  Endpoint M-Value (n=228, n=231) | 26.27 (7.41) | 27.99 (7.28)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.776, ANOVA — P-value for Baseline MODD; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.02, 95% CI [-0.14 to 0.19] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.737, ANOVA — P-value for Baseline M-Value; ANOVA Model: Variable=Treatment + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 1.27, 95% CI [-6.14 to 8.68] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.701, ANCOVA — P-value for 12 Week MODD; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.03, 95% CI [-0.19 to 0.13] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.400, ANCOVA — P-value for 12 Week M-Value; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 1.58, 95% CI [-2.11 to 5.27] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.321, ANCOVA — P-value for 24 Week MODD; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.09, 95% CI [-0.26 to 0.09] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.179, ANCOVA — P-value for 24 Week M-Value; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 2.52, 95% CI [-1.16 to 6.21] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.573, ANCOVA — P-value for 36 Week MODD; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.05, 95% CI [-0.22 to 0.12] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.629, ANCOVA — P-value for 36 Week M-Value; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.95, 95% CI [-4.79 to 2.90] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.250, ANCOVA — P-value for Endpoint MODD. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -0.09, 95% CI [-0.26 to 0.07] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.362, ANCOVA — P-value for Endpoint M-Value; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = -1.72, 95% CI [-5.44 to 1.99] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Number of Patients With at Least One Self-reported Hypoglycemic Episode, Including Nocturnal (and Non-nocturnal) Hypoglycemia
Description: Hypoglycemic episode defined: any time patient felt that he/she was experiencing a sign or symptom associated with hypoglycemia, or had old Roche blood glucose level <70 mg/dL even if not associated with signs, symptoms, or treatment consistent with current guidelines. Nocturnal hypoglycemia defined: any hypoglycemic event that occurred between bedtime and waking. Non-nocturnal hypoglycemia defined: any hypoglycemic event that occurred between waking and bedtime. Overall episodes: those that occurred at any time during the post-randomization visits. Endpoint: last visit interval based on LOCF.
Time Frame: Baseline to 36 Weeks
Population: Number of randomized patients with baseline and at least one post-baseline value. Intent to treat population. The last visit of trial interval was used to calculate hypoglycemic episodes at Endpoint if patient completes trial and last observation carried forward was used if the patient dropped out of the study early.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
participants
  Endpoint Hypoglycemic Episodes | 87 | 106
  Overall Hypoglycemic Episodes | 178 | 179
  Endpoint Nocturnal Hypoglycemic Episodes | 30 | 37
  Overall Nocturnal Hypoglycemic Episodes | 112 | 112
  Endpoint Non-Nocturnal Hypoglycemic Episodes | 71 | 98
  Overall Non-Nocturnal Hypoglycemic Episodes | 175 | 179
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.094, Fisher Exact — P-value for Endpoint Hypoglycemic Episodes
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 1.00, Fisher Exact — P-value for Overall Hypoglycemic Episodes
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.430, Fisher Exact — P-value for Endpoint Nocturnal Hypoglycemic Episodes
Statistical Analysis 4: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 1.00, Fisher Exact — P-value for Overall Nocturnal Hypoglycemic Episodes
Statistical Analysis 5: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.013, Fisher Exact — P-value for Endpoint Non-Nocturnal Hypoglycemic Episodes
Statistical Analysis 6: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.756, Fisher Exact — P-value for Overall Non-Nocturnal Hypoglycemic Episodes

7. Secondary Outcome: 30-Day Adjusted Rates of Self-Reported Hypoglycemic Episodes (Including Nocturnal and Non-Nocturnal)
Description: as for outcome 6
Time Frame: Baseline to 36 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hypoglycemic event per 30 days
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
hypoglycemic event per 30 days
  Endpoint Hypoglycemic Rate | 1.57 (2.98) | 2.19 (3.60)
  Overall Hypoglycemic Rate | 1.88 (2.44) | 2.21 (2.87)
  Endpoint Nocturnal Hypoglycemic Rate | 0.26 (0.79) | 0.32 (0.84)
  Overall Nocturnal Hypoglycemic Rate | 0.26 (0.43) | 0.28 (0.50)
  Endpoint Non-Nocturnal Hypoglycemic Rate | 1.31 (2.80) | 1.87 (3.29)
  Overall Non-Nocturnal Hypoglycemic Rate | 1.63 (2.25) | 1.93 (2.71)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.022, ANOVA — P-value for Endpoint Hypoglycemic Rate; ANOVA Model: Rank of Variable = Treatment + Sufonylurea Stratum + Country + Baseline HbA1c Stratum
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.218, ANOVA — P-value for Overall Hypoglycemic Rate; ANOVA Model: Rank of Variable = Treatment + Sufonylurea Stratum + Country + Baseline HbA1c Stratum
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.311, ANOVA — P-value for Endpoint Nocturnal Hypoglycemic Rate; ANOVA Model: Rank of Variable = Treatment + Sufonylurea Stratum + Country + Baseline HbA1c Stratum
Statistical Analysis 4: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.615, ANOVA — P-value for Overall Nocturnal Hypoglycemic Rate; ANOVA Model: Rank of Variable = Treatment + Sufonylurea Stratum + Country + Baseline HbA1c Stratum
Statistical Analysis 5: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.018, ANOVA — P-value for Endpoint Non-Nocturnal Hypoglycemic Rate; ANOVA Model: Rank of Variable = Treatment + Sufonylurea Stratum + Country + Baseline HbA1c Stratum
Statistical Analysis 6: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.255, ANOVA — P-value for Overall Non-Nocturnal Hypoglycemic Rate; ANOVA Model: Rank of Variable = Treatment + Sufonylurea Stratum + Country + Baseline HbA1c Stratum

8. Secondary Outcome: Number of Patients With at Least One Severe Hypoglycemia Episode
Description: Severe hypoglycemia was defined as hypoglycemic event that meets at least one of the following criteria: not capable of treating self and blood glucose <2.8 millimoles per liter (mmol/L); not capable of treating self, blood glucose is missing and prompt recovery after oral carbohydrate or glucagon or intravenous glucose; hypoglycemic event outcome was coma, hopitalization, emergency room visit, or automobile accident. The overall category is a severe hypoglycemic event that occurred at any time during the post-randomization visits. Endpoint: last visit interval based on LOCF.
Time Frame: Baseline to 36 Weeks
Population: Number of randomized patients with baseline and at least one post-baseline value. Intent to treat population. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
participants
  Endpoint Severe Hypoglycemic Episodes | 1 | 1
  Overall Severe Hypoglycemic Episodes | 8 | 5
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.416, Fisher Exact — P-value for Overall Severe Hypoglycemic Episodes

9. Secondary Outcome: Endpoint Insulin Dose Per Body Weight; Total, Basal, and Prandial
Description: Total daily insulin dose adjusted for body weight (Units of insulin per kilogram per day [U/kg/day]) was assessed. Basal insulin is the amount of insulin required to manage normal daily blood glucose fluctuations. Prandial insulin is taken at meal time. Insulin glargine is a basal insulin and insulin lispro is a prandial insulin. Insulin lispro mid-mix is a 50/50 mixture of a basal insulin and insulin lispro. Endpoint: last visit interval based on LOCF.
Time Frame: 36 Weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: U/kg/day
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
U/kg/day
  Daily Basal (n=239, n=240) | 0.27 (0.07) | 0.35 (0.07)
  Daily Prandial (n=239, n=130) | 0.36 (0.08) | 0.29 (0.08)
  Daily Total (n=239, n=240) | 0.57 (0.11) | 0.51 (0.11)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Daily Basal; ANCOVA Model: Variable=Treatment + Country + Baseline HbA1c stratum + Sulfonylurea stratum; Mean Difference (Net) = -0.08, 95% CI [-0.12 to -0.05] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Daily Prandial; ANCOVA Model: Variable=Treatment + Country + Baseline HbA1c stratum + Sulfonylurea stratum; Mean Difference (Net) = 0.07, 95% CI [0.04 to 0.11] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value for Daily Total; ANCOVA Model: Variable=Treatment + Country + Baseline HbA1c stratum + Sulfonylurea stratum; Mean Difference (Net) = 0.07, 95% CI [0.01 to 0.12] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Endpoint Insulin Dose; Total, Basal, and Prandial
Description: Total daily insulin dose (Units of insulin per day [U/day]) was assessed. Basal insulin is the amount of insulin required to manage normal daily blood glucose fluctuations. Prandial insulin is taken at meal time. Insulin glargine is a basal insulin and insulin lispro is a prandial insulin. Insulin lispro mid-mix is a 50/50 mixture of a basal insulin and insulin lispro. Endpoint: last visit interval based on LOCF.
Time Frame: 36 Weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: U/day
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
U/day
  Daily Basal (n=239, n=240) | 19.90 (5.46) | 26.86 (5.37)
  Daily Prandial (n=239, n=130) | 27.73 (6.23) | 21.68 (6.19)
  Daily Total (n=239, n=240) | 43.44 (8.65) | 38.25 (8.51)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Daily Basal; ANCOVA Model: Variable=Treatment + Country + Baseline HbA1c stratum + Sulfonylurea stratum; Mean Difference (Net) = -6.96, 95% CI [-9.65 to -4.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Daily Prandial; ANCOVA Model: Variable=Treatment + Country + Baseline HbA1c stratum + Sulfonylurea stratum; Mean Difference (Net) = 6.05, 95% CI [3.39 to 8.71] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value for Daily Total; ANCOVA Model: Variable=Treatment + Country + Baseline HbA1c stratum + Sulfonylurea stratum; Mean Difference (Net) = 5.20, 95% CI [0.93 to 9.46] — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: Number of Insulin Injections Per Day
Time Frame: Weeks 12, 24, 30, 36
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: insulin injections
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
insulin injections
  Week 12 | 1.33 (0.19) | 1.00 (0.18)
  Week 24 | 1.97 (0.28) | 1.76 (0.27)
  Week 30 | 2.05 (0.30) | 1.81 (0.30)
  Week 36 | 2.03 (0.30) | 1.80 (0.29)
  Endpoint | 1.98 (0.30) | 1.79 (0.29)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Week 12; ANCOVA Model: Variable=Treatment + Baseline HbA1c stratum + Sulfonylurea stratum + Country; Mean Difference (Net) = 0.33, 95% CI [0.24 to 0.42] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Week 24; ANCOVA Model: Variable=Treatment + Baseline HbA1c stratum + Sulfonylurea stratum + Country; Mean Difference (Net) = 0.22, 95% CI [0.07 to 0.36] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Week 30; ANCOVA Model: Variable=Treatment + Baseline + Baseline HbA1c stratum + Country + Sulfonylurea stratum; Mean Difference (Net) = 0.24, 95% CI [0.09 to 0.40] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value for Week 36; ANCOVA Model: Variable=Treatment + Baseline HbA1c stratum + Sulfonylurea stratum + Country; Mean Difference (Net) = 0.22, 95% CI [0.07 to 0.38] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.011, ANCOVA — P-value for Endpoint. (last observation carried forward); ANCOVA Model: Variable=Treatment + Baseline HbA1c stratum + Sulfonylurea stratum + Country; Mean Difference (Net) = 0.19, 95% CI [0.04 to 0.34] — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Change From Baseline in Absolute Body Weight at 36 Week Endpoint
Description: Change in body weight was calculated as weight at endpoint (last observation carried forward) minus weight at baseline.
Time Frame: Baseline, 36 Weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Number analyzed (Participants) | 239 | 240
kilograms
  Baseline | 76.71 (5.09) | 77.00 (5.01)
  Change from Baseline | 3.09 (1.44) | 3.19 (1.42)
Statistical Analysis 1: Comparison: Insulin Lispro Mid Mixture vs Insulin Glargine; Test type: Superiority or Other; p = 0.803, ANCOVA — P-value for Change from Baseline; ANCOVA Model: Variable=Treatment + Baseline + Sulfonylurea stratum + Country + Baseline HbA1c stratum; Mean Difference (Net) = -0.09, 95% CI [-0.80 to 0.62] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Arm/Group | Insulin Lispro Mid Mixture | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 11/239 | 11/240
Other Adverse Events (participants affected / at risk) | 91/239 | 92/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro Mid Mixture (N=239) | Insulin Glargine (N=240)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) — Death (insulin glargine patient)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Death (insulin glargine patient)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro Mid Mixture (N=239) | Insulin Glargine (N=240)
Cataract (Eye disorders) | 0 (0) | 3 (4)
Diabetic retinopathy (Eye disorders) | 1 (1) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 8 (9)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Fatigue (General disorders) | 4 (5) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 4 (7) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6) | 12 (12)
Gastroenteritis (Infections and infestations) | 3 (4) | 3 (3)
Influenza (Infections and infestations) | 3 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 20 (31) | 21 (22)
Upper respiratory tract infection (Infections and infestations) | 4 (7) | 6 (6)
Urinary tract infection (Infections and infestations) | 5 (5) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 2 (3)
Headache (Nervous system disorders) | 4 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days